CLINICAL TRIAL: NCT05589701
Title: Prospective Registry Trail COMparing Stereotactic Body Radiotherpy (SBRT) to Conventional PAlliative RadioTherapy (CRT) in Patients With Spinal Metastases
Brief Title: Comparing SBRT to CRT in Patients With Spinal Metastases
Acronym: COMBAT
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5085
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Spinal Metastases
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stereotactic Radiotherapy (SBRT): Standard of care stereotactic radiotherapy.
  Interventions: Radiation: Radiotherapy
- Conventional Radiotherapy (CRT): Standard of care conventional radiotherapy.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Standard of care radiotherapy administered as per institutional guidelines.

SUMMARY:
This is a single institutional registry-based, prospective, observational study to describe radiation oncologists' decision making during evaluation of patients and to compare real-world outcomes of SBRT vs CRT.

A registry-based trial involves observing the effect of something without manipulating it.

DETAILED DESCRIPTION:
The purpose of this study is to study the differences between CRT and SBRT. The investigator's are assessing radiation oncologists' decision-making during the evaluation of patients with spinal metastases by requesting radiation oncologists complete a questionnaire. Additionally, the investigator's will compare outcomes, including local progression, pain response and overall survival between SBRT and CRT. By collecting this information, the investigator's will develop an evidence-based algorithm that may be used to support medical decision-making for others with spinal metastases in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Patients seen at the Princess Margaret Cancer Centre with painful spinal metastases amenable to radiation treatment.
* Confirmation of diagnosis: a) Known/documented prior histological cancer diagnosis
* Able to provide written consent
* ECOG performance status 0-3

Exclusion Criteria:

* Prior radiotherapy, with fields overlapping, resulting in excessive doses to organs at risk
* Lymphoma, myeloma or germ cell malignancies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have MRI- or CT-documented spinal metastases and are suitable for receiving radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Describe physician decision-making when making a recommendation for SBRT vs CRT in spine metastasis patients requiring radiation. | 2 years
  Physician's decision making will be assessed by a questionnaire containing 6 questions, including questions on variations of practice and the role of a number of factors that may influence a physician's recommendation for spine metastasis patients requiring radiation (SBRT vs CRT).

SECONDARY OUTCOMES:
Assess local progression free survival. | 2 years
  Based on available imaging, compare local progression free survival outcomes of patients treated with SBRT vs CRT.
Measure pain response | 2 years
  Using a patient reported scale (0 (no pain) to 10 (worst pain imaginable)), compare pain outcomes of patients treated with SBRT vs CRT.
Assess adverse events | 2 years
  Compare adverse events, collected through standard of care follow up, which occur for patients treated with SBRT vs CRT.
Measure overall survival | 2 years
  Compare overall survival, collected through medical records, for patients treated with SBRT vs CRT.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada